CLINICAL TRIAL: NCT05144633
Title: Blue Protocol and Eko Artificial Intelligence Are Best (BEA-BEST)
Acronym: BEA-BEST
Status: Recruiting | Type: Observational
Sponsor: University of Louisville (Other)
Collaborators: Eko Devices, Inc. (Industry)
Responsible Party: Principal Investigator, Rodrigo Cavallazzi, MD, Associate Professor of Medicine, University of Louisville
Other Study IDs: 21.0389
Record Dates: First submitted 2021-08-01; First posted 2021-12-03 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-06

CONDITIONS: Acute Respiratory Failure
MeSH Terms: interventions — Auscultation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Acute Respiratory failure: Patients presenting to the Emergency Department in acute respiratory failure. These patients may or may not have a diagnosis of chronic lung disease.
  Interventions: Device: Auscultation

INTERVENTIONS:
Device: Auscultation — This study will be to determine if the addition of Eko AI-assisted lung auscultation examination to a standard of care Pulmonary POCUS + assists with acute respiratory failure diagnosis.

SUMMARY:
This is an observational study that will be enrolling University of Louisville patients who present to the Emergency Department in Acute Respiratory Failure. This study will be to determine if the addition of Eko AI-assisted lung auscultation examination to a standard of care Pulmonary POCUS + assists with acute respiratory failure diagnosis.

DETAILED DESCRIPTION:
Once identified and consented, the subject will undergo both POCUS and AI-assisted lung auscultation using an Eko CORE stethoscope. The POCUS protocol described here is the standard of care for patients who present in acute respiratory failure to the Emergency Room and both groups will receive this standardized care during the study.

Upon hospital discharge, the final discharge diagnosis will be used as the ground truth for assessing the accuracy of the POCUS protocol. The POCUS exam and the EkoAI exam may be performed wherever the subject is located in the hospital when first enrolled in the study. If possible, both exams should be performed immediately, in either order. They will be performed by the same examiner.

Both the POCUS and the EkoAI exam will be analysed by an investigator blinded to the final diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older presenting to the ED or admitted to the hospital within 12 hours of enrollment
* Acute respiratory failure defined as new onset shortness of breath initiated within the last 7 days, and new or increasing need for oxygen therapy
* The patient or patient's legal health care proxy consents to participation

Exclusion Criteria:

Unwillingness to consent

* Patients with trauma as the cause of ARF
* Patients with pneumothorax as the cause of ARF
* Inability to perform pulmonary POCUS or lung auscultation (e.g. dressing on the chest)
* Unwilling or unable to complete the minimum of 12 lung sound stethoscope recordings.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18years and older, presenting to the Emergency Department in acute respiratory failure.
  These patients may or may not have a diagnosis of chronic lung disease. It may be necessary to enroll more than 100 subjects in order to achieve 100 completed datasets.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Measure the accuracy of POCUS for the diagnosis of acute respiratory failure | 2 years
  POCUS consists of an ultrasound examination at bedside. We will perform lung ultrasound and the pattern of lung ultrasound will be used to diagnose the cause of acute respiratory failure. The reference standard will be the the final diagnosis by the clinician. The accuracy measures will include sensitivity, specificity, positive predictive value, and negative predictive value.
Measure the accuracy of POCUS plus Eko for the diagnosis of acute respiratory failure. AI-assisted lung auscultation for the diagnosis of the case of acute respiratory failure. | 2 years
  POCUS was described above. Ekos consists of a digital stethoscope. The lung auscultation pattern will be used to determine the cause of acute respiratory failure. POCUS and Eko will be integrated to establish the cause of acute respiratory failure. The reference standard will be the final diagnosis by the clinician.
Agreement between POCUS and Eko CORE | 2 years
  We will measure Kappa statistic.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Cavallazzi, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No